CLINICAL TRIAL: NCT01963442
Title: A Non-Inferiority, Multicentered, Controlled, Randomized, Double Blinded Study Investigating the Antibiotic Treatment Duration (3-day Versus 8-day) for Subjects Admitted to Emergency Services With Acute Non-severe Community Acquired Pneumonia (CAP)
Brief Title: Short Duration Treatment of Non-severe Community Acquired Pneumonia
Acronym: PTC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Anne-claude Cremieux, Clinical Coordinator, Versailles Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PHRC-12-202.0496 - PTC; 2013-000265-36 (EudraCT Number)
Record Dates: First submitted 2013-10-09; First posted 2013-10-16 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Community Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — X-Rays; Blood Specimen Collection; Cell Count; C-Reactive Protein; Amoxicillin-Potassium Clavulanate Combination; beta-Lactams

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amoxicillin/Clavulanic acid treatment (Active Comparator): after 3 day treatment of β-lactams, the subjects receive 5-day treatment of Amoxicillin/clavulanic acid. Chest X-ray performed at admission and Day 30 and replapses. 'blood sampling /Cell Counts/CRP/Biochemistry' performed at Day 0, Day 30 and relapse
  Interventions: Radiation: Chest X-ray; Biological: blood sampling /Cell Counts/ C reactive protein (CRP)/Biochemistry; Drug: Augmentin; Drug: Beta-Lactams
- placebo treatment (Placebo Comparator): after 3-day treatment of β-lactams, the subjects receive 5-day treatment of placebo. Chest X-ray performed at admission and Day 30 and replapse. blood sampling /Cell Counts/CRP/Biochemistry' performed at Day 0, Day 30 and relapse
  Interventions: Radiation: Chest X-ray; Biological: blood sampling /Cell Counts/ C reactive protein (CRP)/Biochemistry; Drug: Placebo (for Augmentin); Drug: Beta-Lactams

INTERVENTIONS:
Radiation: Chest X-ray — at Day 0, Day 30 and relapse
Biological: blood sampling /Cell Counts/ C reactive protein (CRP)/Biochemistry
Drug: Augmentin — 2 tablets 3 times a day for 5 days from Day 3
  Arms: Amoxicillin/Clavulanic acid treatment
Drug: Placebo (for Augmentin) — 2 tablets 3 times a day for 5 days from Day 3
  Arms: placebo treatment
Drug: Beta-Lactams — administered from Day 0 to Day 3

SUMMARY:
To investigate the non inferiority of a short lasting antibiotic treatment (3 days) when compared to a long lasting antibiotic treatment (8 days), at Day 15 after the beginning of treatment in terms of clinical efficacy, in adults admitted to emergency services for a non severe Community Acquired Pneumonia (PAC), who responded well to 3 days of beta-lactamin treatment (3GC or A/AC).

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years old or over.
* admitted three days before for Community Acquired Pneumonia (CAP) defined by at least one clinical sign of pneumonia (dyspnea, cough, mucopurulent sputum, crackling sound on lungs) associated with a temperature >38°C on admission, and a new infiltrate consistent with pneumonia on chest x-ray, who responded favorably to 3 days of treatment with β-lactams (third generation injectable cephalosporin or amoxicillin-clavulanate)
* able to take oral medication.
* has given its informed consent.

Exclusion Criteria:

* Creatinin < 30ml/min
* History of jaundice / hepatic impairment associated with amoxicillin / clavulanic acid
* History of hypersensitivity to beta-lactam
* Presence of complications or severity of pneumonia (abscess , significant pleural effusion, severe chronic respiratory failure , septic shock, respiratory condition requiring the passage resuscitation).
* Known immunocompromised terrain ( asplenia , neutropenia, agammaglobulinemia , immunosuppressants, graft corticosteroids , myeloma , lymphoma, known HIV , sickle cell anemia , CHILD C cirrhosis).
* Antibiotic treatment exceeding 24 hours prior admission.
* Suspected atypical bacteria requiring combined antibiotics therapy .(Subjects who received a single dose of macrolides or fluoroquinolones emergency will not be excluded) .
* Legionella suspected on clinical, biological and radiological criteria .
* Subjects with clinical or epidemiological environment leading to suspect a healthcare-associated pneumonia with antibiotic resistant pathogen.
* Suspicion of pneumonia by aspiration.
* Intercurrent infection requiring antibiotic treatment.
* Pregnant women .
* Breastfeeding .
* Allergy to antibiotics in use.
* Life expectancy <1 month .
* Subject without health insurance.
* Subjects without home adress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2013-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
clinical evaluation at Day 15 | Day 15
  Clinical evaluation at Day 15 composed of the composite measure of the Clinical examination for clinical symptoms of CAP, recording of the body temperature and confirmation that no additionnal antibiotic treatment was required from Day 8

SECONDARY OUTCOMES:
clinical evaluation at Day 30 | Day 30
  Clinical evaluation at Day 30 composed of the composite measure of the Clinical examination for clinical symptoms of CAP, recording of the body temperature and Evaluation of replapse or aggravation of pneumonia or any other respiratory infections in subjects considered cured at Day 15.

OTHER OUTCOMES:
mortality all causes at Day 30 | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Claude CREMIEUX, Pr, Principal Investigator — Central Hospital Raymon Poincaré; Marie Christine DOMBRET, Dr, Principal Investigator — CHU Bichat; Matthieu GROH, Dr, Principal Investigator — CHU Cochin; Elizabeth ROUVEIX, Pr, Principal Investigator — CHU Ambroise Paré; Pascale LONGUET, Dr, Principal Investigator — CH Argenteuil; Daniel BENHAMOU, Dr, Principal Investigator — CHU Rouen; Sylvain DIAMANTIS, Dr, Principal Investigator — Melun Hospital; Jean-Emmanuel Kahn, Dr, Principal Investigator — Foch Hospital; Jean-François BOITIAUX, Dr, Principal Investigator — Pontoise Hospital; Jean-Pierre BEDOS, Pr, Principal Investigator — Central Hospital of Versailles; Jêrome PACANOWSKI, Dr, Principal Investigator — CHU Saint Antoine (Paris); Valérie GARRAIT, Dr, Principal Investigator — CHI CRETEIL; Elena FOIS, Dr, Principal Investigator — CH Saint Denis; Benjamin WYPLOSZ, Pr, Principal Investigator — CH Bicêtre; Véronique DELCEY, Dr, Principal Investigator — CH Lariboisière; Gilles PIALOUX, Dr, Principal Investigator — CH Tenon; Matthieu REVEST, Dr, Principal Investigator — CHU Rennes Pontchaillou; Jean Paul STAHL, Dr, Principal Investigator — University Hospital, Grenoble; Virginie VITRAT, Dr, Principal Investigator — CH Annecy Genevois; Victoire De Lastours, Dr, Principal Investigator — CH Beaujon
Locations (20):
- France (20):
  - CH Argenteuil, Argenteuil
  - CHU Ambroise Paré, Boulogne-Billancourt
  - CH Beaujon, Clichy
  - CHI Creteil, Créteil
  - Central Hospital Raymon Poincaré, Garches
  - CHU de Grenoble, La Tronche
  - CH Versailles, Le Chesnay
  - CH Bicêtre, Le Kremlin Bicètre
  - Melun Hospital, Melun
  - CH d'Annecy Genevois, Metz-Tessy
  - CH Lariboisière, Paris
  - CHU Saint Antoine, Paris
  - CHU Cochin, Paris
  - CHU Bichat, Paris
  - CH Tenon, Paris
  - CH Pontoise, Pontoise
  - CHU Rennes Pontchaillou, Rennes
  - CHU Rouen, Rouen
  - CH Saint Denis, Saint-Denis
  - Foch Hospital, Suresnes

REFERENCES:
- [Derived] Dinh A, Duran C, Ropers J, Bouchand F, Deconinck L, Matt M, Senard O, Lagrange A, Mellon G, Calin R, Makhloufi S, de Lastours V, Mathieu E, Kahn JE, Rouveix E, Grenet J, Dumoulin J, Chinet T, Pepin M, Delcey V, Diamantis S, Benhamou D, Vitrat V, Dombret MC, Renaud B, Claessens YE, Labarere J, Bedos JP, Aegerter P, Cremieux AC; Pneumonia short treatment (PTC) study group. Exclusive oral antibiotic treatment for hospitalized community-acquired pneumonia: a post-hoc analysis of a randomized clinical trial. Clin Microbiol Infect. 2024 Aug;30(8):1020-1028. doi: 10.1016/j.cmi.2024.05.003. Epub 2024 May 9. PMID 38734138
- [Derived] Dinh A, Ropers J, Duran C, Davido B, Deconinck L, Matt M, Senard O, Lagrange A, Makhloufi S, Mellon G, de Lastours V, Bouchand F, Mathieu E, Kahn JE, Rouveix E, Grenet J, Dumoulin J, Chinet T, Pepin M, Delcey V, Diamantis S, Benhamou D, Vitrat V, Dombret MC, Renaud B, Perronne C, Claessens YE, Labarere J, Bedos JP, Aegerter P, Cremieux AC; Pneumonia Short Treatment (PTC) Study Group. Discontinuing beta-lactam treatment after 3 days for patients with community-acquired pneumonia in non-critical care wards (PTC): a double-blind, randomised, placebo-controlled, non-inferiority trial. Lancet. 2021 Mar 27;397(10280):1195-1203. doi: 10.1016/S0140-6736(21)00313-5. PMID 33773631